CLINICAL TRIAL: NCT04108442
Title: Patient Satisfaction With Virtual Postoperative Visit
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 19-00549
Record Dates: First submitted 2019-08-22; First posted 2019-09-30 (Actual); Last update posted 2020-10-09 (Actual); Status verified 2020-10

CONDITIONS: Post-Op Complication
MeSH Terms: conditions — Postoperative Complications

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Traditional (Active Comparator)
  Interventions: Behavioral: Traditional
- Virtual (Experimental)
  Interventions: Behavioral: Virtual

INTERVENTIONS:
Behavioral: Traditional — Surgeons (rather than individual subjects) will be randomized to traditional Postoperative follow-up modality groups. They will adhere to this form of postoperative follow-up for all of their surgical patients (subjects) for one month.
  Arms: Traditional
Behavioral: Virtual — Surgeons (rather than individual subjects) will be randomized to virtual postoperative follow-up modality group. They will adhere to that form of postoperative follow-up for all of their surgical patients (subjects) for one month.
  Arms: Virtual

SUMMARY:
This is a prospective, randomized study designed to evaluate the effects of different initial postoperative follow-up modalities. Given the nature of the study, it is not possible for either the surgeons or the subjects to be blinded. To reduce bias that may occur due to each surgeon's personal preference for postoperative follow-up modality, the surgeons (rather than individual subjects) will be randomized to one of two postoperative follow-up modality groups (traditional or virtual).

ELIGIBILITY:
Inclusion Criteria:

* > 18 years old
* < 60 years old
* Undergoing knee arthroscopy procedure

Exclusion Criteria:

* < 18 years old
* > 60 years old

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 122 (Actual)
Dates: Start 2019-08-01 (Actual); Primary Completion 2020-03-01 (Actual); Study Completion 2020-03-01 (Actual)

PRIMARY OUTCOMES:
Patient Satisfaction with their surgeon | 6 Months
  Patients will report their satisfaction with their surgical experience 6 weeks after surgery using a 10-point Likert scale, 0-"Completely Dissatisfied, 10-"Completely Satisfied"

CONTACTS AND LOCATIONS:
Overall Officials: Kirk Campbell, MD, Principal Investigator — New York Langone Health
Locations (1):
- NYU Langone Health, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in this article, after deidentification (text, tables, figures, and appendices).
Supporting Information: Study Protocol, SAP
Time Frame: Beginning 9 months and ending 36 months following article publication or as required by a condition of awards and agreements supporting the research.
Access Criteria: The investigator who proposed to use the data.